CLINICAL TRIAL: NCT00878436
Title: Phase I/II Randomized Trial of LBH589 (Panobinostat) at Two Dose Levels Combined With Bicalutamide (Casodex) in Men With Castration-resistant Prostate Cancer
Brief Title: Safety and Efficacy Studies of Panobinostat and Bicalutamide in Patients With Recurrent Prostate Cancer After Castration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-479
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: histone deacetylase inhibitor; hormone therapy; androgen-independent; PSA; androgen receptor
MeSH Terms: conditions — Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — Panobinostat; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (120 mg/week) (Experimental): Each treatment cycle has 21 days:
  Bicalutamide (Casodex®) 50mg P.O. daily, continuously, with the addition of:
  40 mg Panobinostat 3 times per week (120 mg per week) for 2 consecutive weeks with one week rest
  Interventions: Drug: Panobinostat; Drug: Bicalutamide
- Arm B (60 mg/week)-Closed to accrual (Experimental): Each treatment cycle has 21 days:
  Bicalutamide (Casodex®) 50mg P.O. daily, continuously, with the addition of:
  20 mg Panobinostat 3 times per week (60 mg per week) for 2 consecutive weeks with one week rest
  Interventions: Drug: Panobinostat; Drug: Bicalutamide

INTERVENTIONS:
Drug: Panobinostat
  Other Names: LBH589
Drug: Bicalutamide
  Other Names: Casodex

SUMMARY:
This trial is designed to investigate the safety, dosing schedule, and efficacy of the combination treatment of Panobinostat (a histone deacetylase inhibitor) and hormone therapy for recurrent prostate cancer. This trial is at its Phase II stage. As of July 23, 2013 Arm B was closed to accrual, all the remaining slots in accrual will be allocated to Arm A.

DETAILED DESCRIPTION:
The preclinical data indicate that Panobinostat restores the sensitivity of androgen-independent cells to bicalutamide (Casodex®) and the combination has synergistic inhibitory activity. Here, we hypothesize that treatment of castration-resistant patients with Panobinostat will enhance the response to the second line hormone therapy with bicalutamide (Casodex®). In the proposed phase I study, the maximum tolerated dose of tri-weekly, intermittent oral Panobinostat at three different dose levels (60, 90, 120 mg/week) in combination with Casodex (50mg PO) will be determined; The following phase II study will evaluated the efficacies of 9-month treatments of the selected Panobinostat-Casodex combination and also a lower dose of Panobinostat. We expect that Casodex-Panobinostat combination treatment of castration-resistant patients will prevent biochemical and/or metastatic disease progression of these patients compared to historical controls in the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Patients must meet laboratory criteria
* Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal.
* ECOG Performance Status of ≤ 2
* Documented history of adenocarcinoma of the prostate.
* Patients must have evidence of disease progression while receiving androgen suppression therapy by orchiectomy or other primary hormonal therapy including, but not limited to (LHRH agonist therapy (e.g., leuprolide or goserelin) or LHRH antagonist (e.g. aberelix). Note: patients who have not undergone bilateral orchiectomy must continue LHRH therapy while on protocol
* Testosterone must be < 50 ng/dl confirmed within 4 weeks prior to registration for patients on LHRH therapy
* Patients must have evidence of disease progression with either one or both of the conditions listed:

  * Biochemical progression only
  * Metastases on bone scan
* Patients may have received one chemotherapy, investigational agent or immunotherapy in the neoadjuvant, adjuvant setting or during initial LHRH therapy with new evidence of disease progression after discontinuation of therapy for ≥ 2 weeks.
* Patients must have received one or more prior second line hormone therapy for progression while on LHRH treatment or orchiectomy.
* Patients treated with one first line chemotherapy combination for hormone refractory progression ≥ 4 weeks prior to registration who have evidence of disease progression and had only one second line hormone therapy and did not experience PSA response to bicalutamide (Casodex®) withdrawal.

Exclusion Criteria:

* Prior treatment with an HDAC inhibitor
* Impaired cardiac function including any one of the following:

  * Screening ECG with a QTc > 450 msec confirmed by central laboratory prior to enrollment to the study
  * Patients with congenital long QT syndrome
  * History of sustained ventricular tachycardia
  * Any history of ventricular fibrillation or torsades de pointes
  * Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
  * Patients with a myocardial infarction or unstable angina within 6 months of study entry
  * Congestive heart failure (NY Heart Association class III or IV)
  * Right bundle branch block in conjunction with left anterior hemi-block (bifasicular block)
* Uncontrolled hypertension
* Concomitant use of drugs with a risk of causing torsades de pointes
* Concomitant use of CYP3A4 inhibitors
* Patients with unresolved diarrhea greater than CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Concomitant use of any anti-cancer therapy or radiation therapy.
* Male patients whose sexual partners are WOCBP not using effective birth control
* Patients with a history of another primary malignancy within the last 2 years that was not curatively treated, excluding basal or squamous cell carcinoma of the skin
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Patients previously treated with bicalutamide (Casodex®) who experienced a PSA withdrawal response in the washout period as described in Inclusion #11 will not be eligible
* Concurrent use of estrogens or estrogen like substances (i.e. PC-SPES, Saw Palmetto, or other herbal product which may contain phytoestrogens) is not allowed. Prior use of these agents will need to be discontinued at least 4 weeks prior to enrollment, for the above.
* Radiotherapy within the 4 weeks prior to registration
* Inadequate bone marrow function measured 28 days prior to registration
* No serious concurrent medical illness or active infection that would jeopardize the ability of the patient to receive therapy as outlined in the protocol with reasonable safety.
* Liver metastasis.
* The use of bisphosphonates in the absence of metastasis will not be allowed. Patients on bisphosphonates for more than 4 weeks for asymptomatic bone metastasis and with continued evidence of PSA progression may continue on bisphosphonates every 4 weeks.
* Hydronephrosis with impaired renal function.
* Active spinal cord compression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ferrari, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - North Shore University Hospital-Monter Cancer Center, Lake Success, New York
  - NYU Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Members of the research team have attempted to contact the PI, unsuccessfully, and are unable to answer questions regarding results.
Groups:
- LBH 40mg: Participants assigned to this arm received 40mg of LBH589 (LBH) three times a week (for a total weekly dose of 120mg). Additionally, they received 50mg of bicalutamide (Bic) daily.
- LBH 20mg: Participants assigned to this arm received 20mg of LBH589 (LBH) three times a week (for a total weekly dose of 60mg). Additionally, they received 50mg of bicalutamide (Bic) daily.
Period: Overall Study
Arm/Group | LBH 40mg | LBH 20mg
Started | 28 | 24
Completed 2 Cycles | 21 | 20
6 Months | 8 | 0
Completed | 5 | 0
Not Completed | 23 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LBH 40mg | LBH 20mg | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Median (Full Range); unit: years] | 69 [48 to 84] | 69 [50 to 83] | 69 [48 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 24 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Free of Progression and Without Symptomatic Deterioration
Description: measured by PSA and /or metastases progression criteria by body CT following RECIST criteria 1.1 and/or bones scan following the appearance of at least 2 new bone metastases and confirmation of 2 additional bone metastasis on a subsequent bone scan 6-8 weeks later and/or clinical progression.
  Only participants who completed two or more treatment cycles were assessed for this outcome measure.
Time Frame: 9 months
Measure: Number; unit: percentage of Participants
Arm/Group | LBH 40mg | LBH 20mg
Number analyzed (Participants) | 21 | 20
percentage of Participants | 24 | 9

2. Primary Outcome: Percentage of Patients Free of Progression and Without Symptomatic Deterioration
Description: as for outcome 1
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | LBH 40mg | LBH 20mg
Number analyzed (Participants) | 21 | 20
percentage of participants | 42 | 19

3. Secondary Outcome: Time to PSA Progression
Description: PSA progression is defined as a 25% or greater increase in PSA and an absolute increase value of 2 ng/ml or more over a nadir or baseline documented and confirmed by a second value three weeks later
Time Frame: up to 2 years
Population: Unable to locate PI for secondary outcome measure results. Data is not available.
Arm/Group | LBH 40mg | LBH 20mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Patients That Achieve a 50% or Greater PSA Decline by 9 Months of Therapy
Description: Unable to locate PI for secondary outcome measure results. Data is not available.
Time Frame: 9 months
Population: Unable to locate PI for secondary outcome measure results. Data is not available.
Arm/Group | LBH 40mg | LBH 20mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | LBH 40mg | LBH 20mg
Serious Adverse Events (participants affected / at risk) | 11/28 | 5/24
Other Adverse Events (participants affected / at risk) | 26/28 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH 40mg (N=28) | LBH 20mg (N=24)
Acute Renal Failure (Renal and urinary disorders) | 1 | 0
Cardiac Asystole (Cardiac disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Cord Compression (Surgical and medical procedures) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Karposi Sarcoma (General disorders) | 0 | 1
Myelodysplasia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pleural Effusion (Surgical and medical procedures) | 0 | 1
Qtc Prolonged (Cardiac disorders) | 1 | 0
Stomach Pain (Gastrointestinal disorders) | 1 | 0
Subarachoid Hemorrhage (Blood and lymphatic system disorders) | 0 | 1
Subdural Hematoma (Blood and lymphatic system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Ulcers (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH 40mg (N=28) | LBH 20mg (N=24)
Albumin (Metabolism and nutrition disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Altered Taste (Gastrointestinal disorders) | 2 | 1
Anc (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 3
Anorexia (Gastrointestinal disorders) | 7 | 2
Anxiety (Psychiatric disorders) | 3 | 1
Back Pain (General disorders) | 2 | 0
Bilateral Lower Extremity Edema (Blood and lymphatic system disorders) | 1 | 0
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 | 0
Bloating / Distention (Gastrointestinal disorders) | 1 | 0
Blotches (Skin and subcutaneous tissue disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Breast Enlargement (Reproductive system and breast disorders) | 0 | 1
Breast Pain (General disorders) | 1 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bruising (Blood and lymphatic system disorders) | 1 | 0
Burning, Foul Smelling Urination (Infections and infestations) | 0 | 1
Change In Taste (Gastrointestinal disorders) | 2 | 0
Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Ck Elevated (Metabolism and nutrition disorders) | 0 | 1
Cold Sore (Skin and subcutaneous tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 6
Cpk (Metabolism and nutrition disorders) | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 1 | 1
Creatinine Increased (Metabolism and nutrition disorders) | 1 | 0
Decreased Albumin (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Gastrointestinal disorders) | 4 | 4
Decreased Bicarbonates (Metabolism and nutrition disorders) | 1 | 1
Decreased Cpk (Metabolism and nutrition disorders) | 1 | 0
Decreased Creatinine (Metabolism and nutrition disorders) | 1 | 0
Decreased Platelets (Blood and lymphatic system disorders) | 1 | 0
Decreased Sodium (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 1
Dental Abscess (Infections and infestations) | 1 | 1
Depression (Psychiatric disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 14 | 6
Distracted/Concentration Impairment (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 1
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Early Satiety (General disorders) | 0 | 1
Edema- Leg (Blood and lymphatic system disorders) | 1 | 0
Edema- Pedal (Blood and lymphatic system disorders) | 1 | 0
Elevated Alkaline Phosphatase (Metabolism and nutrition disorders) | 0 | 1
Elevated Bun (Metabolism and nutrition disorders) | 0 | 1
Elevated Creatinine (Metabolism and nutrition disorders) | 1 | 2
Elevated Qtc (Cardiac disorders) | 1 | 0
Enlarged L Neck Node (Bl) (Blood and lymphatic system disorders) | 1 | 0
Epigastric Pain (General disorders) | 1 | 0
Facial Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 14 | 16
Flatulence (Gastrointestinal disorders) | 1 | 1
Flu Like Symptoms (General disorders) | 0 | 1
Fracture Right Heel (Injury, poisoning and procedural complications) | 1 | 0
Generalized Aches (General disorders) | 0 | 1
Gerd (Gastrointestinal disorders) | 1 | 0
Gfr (Metabolism and nutrition disorders) | 1 | 1
Hair Loss (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (General disorders) | 3 | 1
Heartburn (Gastrointestinal disorders) | 1 | 2
Hematoma (Skin and subcutaneous tissue disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 3 | 1
Hot Flashes (Endocrine disorders) | 0 | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesmia (Metabolism and nutrition disorders) | 1 | 1
Hypertryglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Imbalance (Ear and labyrinth disorders) | 1 | 1
Increased Creatinine (Metabolism and nutrition disorders) | 3 | 2
Increased Dyspepsia (Gastrointestinal disorders) | 0 | 1
Increased Fatigue (General disorders) | 1 | 0
Increased Ldh (Metabolism and nutrition disorders) | 1 | 0
Increased Nausea (Gastrointestinal disorders) | 1 | 0
Increased Tsh (Endocrine disorders) | 0 | 1
Infection- It. Pylori (Infections and infestations) | 1 | 0
L Eye Conjunctival Hemorrhage (Blood and lymphatic system disorders) | 1 | 0
L Hip Pain From Fall (Injury, poisoning and procedural complications) | 0 | 1
Left Jaw Pain (General disorders) | 1 | 0
Left Sciatic Pain (General disorders) | 0 | 1
Left Scleral Hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Leg Edema (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Light Headed (Nervous system disorders) | 0 | 2
Little Shakey (Musculoskeletal and connective tissue disorders) | 0 | 1
Loose Stools (Gastrointestinal disorders) | 1 | 0
Loss Of Appetite (Gastrointestinal disorders) | 1 | 0
Low Back Pain (General disorders) | 0 | 1
Low Blood Pressure (Cardiac disorders) | 1 | 0
Low Phosphorus (Metabolism and nutrition disorders) | 1 | 0
Low Platelets (Blood and lymphatic system disorders) | 1 | 0
Lower Extremity Edema (Blood and lymphatic system disorders) | 1 | 0
Metallic Taste (Gastrointestinal disorders) | 1 | 0
Mild Nausea (Gastrointestinal disorders) | 0 | 1
Mood Changes (Psychiatric disorders) | 0 | 1
Mucositis- Oral Cavity (Gastrointestinal disorders) | 1 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 1 | 1
Nasal Stuffiness (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 13 | 9
Neck Pain (Gastrointestinal disorders) | 0 | 1
Neuropathy (Bl) (Nervous system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0
Night Sweats (General disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Nose Bleeds (Blood and lymphatic system disorders) | 1 | 0
Occipital Pain (Eye disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Pain, Intermittent (General disorders) | 0 | 1
Petechial Rash (Arms & Legs) (Blood and lymphatic system disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 1 | 0
Platelets Decreased (Blood and lymphatic system disorders) | 1 | 0
R Upper Chest Anular Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rear Pelvic Left Hip Pain (General disorders) | 0 | 1
Rib Pain (General disorders) | 0 | 1
Right Flank Bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Sacral Pain, Intermittent (General disorders) | 0 | 1
Severe Fatigue (General disorders) | 0 | 1
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shoulder Pain (General disorders) | 0 | 1
Sinus Congestion (General disorders) | 1 | 0
Skin Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1
Skin Infection Llq (Infections and infestations) | 0 | 1
Stomach Cramp (Gastrointestinal disorders) | 2 | 0
Sweating (General disorders) | 1 | 0
Swelling Leg (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Taste Changes (Gastrointestinal disorders) | 3 | 0
Tenesmus (Gastrointestinal disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 9
Tinniyus (Ear and labyrinth disorders) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 3 | 1
Urinary Frequency (Renal and urinary disorders) | 1 | 2
Urinary Incontinence (Bl) (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Vasovagal Syncope (Cardiac disorders) | 1 | 0
Ventral Hernia (Musculoskeletal and connective tissue disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Vomiting (1 Episode) (Gastrointestinal disorders) | 1 | 0
Vomitting, Occasion (Gastrointestinal disorders) | 1 | 0
Weak Finger Nails (Skin and subcutaneous tissue disorders) | 0 | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Weight Loss (General disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No